CLINICAL TRIAL: NCT04858165
Title: A Logical Framework for Tailor-made Paradigm Shift Hospital Foodservice to Prevent Malnutrition Among Geriatric Patients in Hospitals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Noraida Binti Omar, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 283284-331068
Record Dates: First submitted 2021-03-30; First posted 2021-04-26 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Hospital Foodservice Satisfaction; Hospital Meals Satisfaction; Elderly, Nutrition, Malnutrition in Elderly, Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (No Intervention): without MY GERYFS
- INTERVENTION (Other): with MY GERYFS
  Interventions: Procedure: MY GERYFS PROTOCOL

INTERVENTIONS:
Procedure: MY GERYFS PROTOCOL — The MY GERYFS will be introduced through a guideline document, dissemination through the department of nursing, notices on the intranet and provision of large signs indicating that MY GERYFS are in progress and the times of meals for each ward. The developed protocol in phase 1 and 2 will be tested in single-centre in a before and after study for its feasibility and safety. In the pre-study, patients will be given usual care. In the post-study, patients will care according to the developed protocol. Clinical outcomes such as malnutrition risk, medical background, anthropometry data, nutrition-focused physical findings, dietary intake, mealtime barrier, Hospital Foodservices satisfaction will be recorded.
  Arms: INTERVENTION

SUMMARY:
Hospital Food service is important for patient recovery by providing necessary aid with adequate meal consumption. Overall, hospital experience can influence patients' satisfaction for the foodservice quality. Thus, it is important to evaluate patient satisfaction with food service to meet consumers' needs in order to prevent malnutrition. The aim of the studies is to develop the Malaysian geriatric patients' hospital foodservice protocol (My GERYFS). There are 3 Phases in this research which is phase 1 is a multicentre cohort study conducted among elderly and healthcare professionals involved in Klang Valley Hospitals. Phase 2 for To develop a tailor-made hospital foodservice protocol for Malaysian geriatric patients with healthcare professional input and phase 3 is to determine the feasibility and cost-effectiveness of MY GERYFS protocol in a Malaysian hospital. Effectiveness of this study protocol can bring benefits to elderly to prevent malnutrition in the hospitals via foodservice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 years and older
* Able to understand and speak Malay or English or both
* Patients who are on oral diet or on Oral Nutrition Support (ONS) or both
* Patients who are admitted for more than 48 hours

Exclusion Criteria:

* Patients who are mentally disturbed
* Critically ill patients
* Patients who are on full enteral or parenteral feeding

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 350 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Nutritional Status | 8 minutes
  Malnutrition assessment of the elderly will be done using Mini Nutritional Assessment-Short Form (MNA-SF). This 7-item questionnaire includes dimensions from food intake, weight status, mobility status, presence of psychological problems and neurological stress level. The total score is categorised into three which are normal nutritional status (12-14 points), at risk of malnutrition (8-11 points) and malnourished (0-7 points).

SECONDARY OUTCOMES:
Medical Background | 5 minutes
  Medical background of the patients will be obtained through patients' medical records and interviewing method. The medical history of the patients includes reasons of admission, date of admission, date of discharge, days of hospitalisation, types and numbers of comorbidities, numbers of drugs prescription, previous hospitalisation and whether the patient has encountered a dietitian visit during hospitalisation. All of these data will be recorded in the self-developed questionnaire.
Anthropometry Measurements | 8 minutes
  Anthropometry measurements of the patients include current and previous body weight, percentage of body weight change, height, body mass index (BMI), mid upper arm circumference (MUAC), calf circumference, triceps skin fold (TSF) and body fat percentage. The body weight of hospitalised patients will be measured using Digital Weighing Scale OMRON HBF-357 and recorded in kilogram (kg) to the nearest 0.1 kg Weight estimation is done to geriatric patients who are unable to stand without assistance or non-ambulatory. The outcome measured will be in Body Mass Index (kg/The Body Mass Index classification will be used as stated in WHO (2004) which is underweight (<18.5kg/m1), normal weight (18.5 to 24.9kg/m2), overweight (25.0 to 29.9kg/m2) and obesity (>30.0kg/m2).
Hand Grip Strength | 2 minutes
  The hand-grip strength test used Jamar Plus+Digital Handgrip Dynamometer as tools of assessment to evaluate muscle strength. The cut-off point recommended for the hadgrip strength is < 26kg/force (men) and <18kg/force (women) consider low strength. While, > 26kg/force (men) and >18kg/force (women) consider normal strength.
Feeding Assistance | 30 seconds
  The respondents' level of feeding assistance will be acquired directly from the patients or caregivers via interviewing method using self-developed questionnaire. The researchers are required to assess the respondents' feeding assistance level during main meals. The level of feeding assistance is classified into four. The level of feeding assistance is classified into dependent, moderate dependent (≥5 minutes), minimal dependent (<5 minutes), and independent.
Visual Ability | 30 seconds
  The respondents' information on visual ability will be acquired via self- reported. The researchers are required to observe if the respondents wear glasses during mealtimes.
Dental Status | 2 minutes
  The dental status will be assessed using Geriatric Oral Health Assessement Index (GOHAI) instrument) 12 questions were developed to evaluate three dimensions of oral health-related quality of life (QoL). These include physical function during eating, psychosocial function including worry or concern about oral health, dissatisfaction with appearance, self-consciousness about oral health an avoidance of social contacts because of oral problems and pain or discomfort including the use of medication to relieve pain or discomfort from the mouth. Each question is given a score 1 to 5. A higher GOHAI score (≥57) indicates better self-reported oral health status and high perception towards oral health, 51 and 56 (average), 12 - 50 (low perception) towards oral health.
Dietary Intake | 10 minutes
  Dietary intake will be obtained by using 24-hour dietary recall for 2 days in the hospital. The dietary intake will be taken among patients who are admitted for ≥ 48 hours and have taken at least two hospital meals. The estimated amount of food will then be converted into grams and later finalised into subject's total energy, macronutrients (protein, carbohydrates and fat) , micronutrients (fat-soluble vitamins, water-soluble vitamins, potassium, sodium, calcium, phosphate, zinc and iron) as well as fibre. The respondents' energy and protein requirements will be estimated above 70% energy and 80% protein consider adequate. This will be done by Nutritionist Pro software.
Mealtime Barriers | 5 minutes
  Mealtime Audit Tool (MAT) instrument is used to measure the respondents' mealtime barriers/issues. This instrument consists of two distinct parts which are Part 1: observation of the time of meal tray arrival (completed by the researcher) and Part 2: list of key challenges or barriers individual patients may experience (completed by the patients). MAT scoring is based on the total of 'NO' responses. The higher the score, the more barriers experienced by the patient.
Hospital Foodservice Satisfaction | 5 minutes
  The Acute Care Hospital Foodservice Patient Satisfaction (ACHFPSQ) questionnaire will be used. Other than that, the statements were grouped into four main dimensions (food quality, meal service quality, staff/service issues, and physical environment) to know the factor scores of the dimensions. The questionnaire uses a 5-point Likert scale (Always = 5, Often = 4, Sometimes = 3, Rarely = 2, and Never =1). This grouping was to measure the highest and lowest score factors affecting satisfaction with hospital foodservice. The relationship between foodservice dimensions with overall satisfaction was assessed with Multiple Linear Regression Analysis. Statements that were worded negatively were scored using the reverse scoring method. The higher the mean score, the better the results were.

CONTACTS AND LOCATIONS:
Locations (5):
- Malaysia (5):
  - Hospital Kuala lumpur, Kuala Lumpur, Kuala Lumpur
  - Hospital Selayang, Batu Caves, Selangor
  - Hospital Tengku Ampuan Rahimah Klang, Klang, Selangor
  - Hospital Pengajar Universiti Putra Malaysia, Serdang, Selangor
  - Hospital Sungai Buloh, Sungai Buloh, Selangor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Omar N, Shafiee SI, Nor'hisham SH, Ibrahim Z, Jamaluddin R, Rahamat S, Mohd Yusof BN, Minhat HS, Sallehuddin H, Mazlan NS. A Logical Framework (MYGERYFS) for Hospital Foodservice to Prevent Malnutrition Among Geriatric Patients in Hospitals, Malaysia: Protocol for a Feasibility Study. JMIR Res Protoc. 2023 Jan 31;12:e42496. doi: 10.2196/42496. PMID 36719732